CLINICAL TRIAL: NCT06295016
Title: Influence of Stressors and Recovery Regulation on the Super-compensation Effect of Endurance Athletes After High-intensity Intensive Training
Brief Title: Stressors and Recovery Regulation on the Super-compensation Effect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: NYCU112130AE
Record Dates: First submitted 2023-11-20; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-11

CONDITIONS: Exercise Overtraining; Stressor, Psychological
Keywords: Supercompensation; High-intensity intensive training; Stressor; Recovery regulation
MeSH Terms: conditions — Overtraining Syndrome; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: The present study is designed as a prospective intervention and prognostic prediction study, employing a single-subject design with a reversal (ABA) design. This design involves a self-controlled intervention experiment with three phases: baseline training period (A), high-intensity, high-volume training period (B), and reduced training period (A). Subsequently, the study aims to explore predictive factors influencing the presence or absence of favorable compensatory training effects following the intervention.
Who Masked: Participant, Investigator
Masking Description: Prior to the commencement of the experiment and during the experimental period, both the participants and the investigator will be unaware of whether the participants exhibit a good response to compensatory training effects. After the participants complete the entire experimental procedure, they will be grouped post hoc based on their outcomes following the intervention, according to predetermined criteria.
  The criteria for determining whether there is a good response to compensatory training effects:
  1. Non-response group: Exercise performance during the tapering period (week 7) shows a significant increase compared to post-intervention (week 6) and is higher than pre-intervention (week 3) exercise performance.
  2. Response group: Exercise performance during the tapering period (week 7) shows a significant increase compared to post-intervention (week 6) and is higher than the change in exercise performance during normal training (= week 3 - week 1).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular training (No Intervention): Participants maintain their regular training habits for 3 weeks.
- High-intensity intensive training (Experimental): Participants increase their regular regular training volume by 10% each week for 3 weeks.
  Interventions: Other: High-intensity intensive training
- Taper (Experimental): Participants gradually reduced to 55% of their regular training volume for 1 week.
  Interventions: Other: Taper

INTERVENTIONS:
Other: High-intensity intensive training — Participants will conduct a 3-weeks of 130% progressive high-intensity intensive training (increasing by 10% each week).
  Week 1: Increase training to 110% of participants' regular training volume. Week 2: Increase training to 120% of participants' regular training volume. Week 3: Increase training to 130% of participants' regular training volume.
  Arms: High-intensity intensive training
Other: Taper — Participants will conduct a 1-week taper phase by gradually reducing to 55% of their regular training volume.
  Day 1: Decrease current training volume by 20%. Day 2: Decrease current training volume by 15%. Day 3: Decrease current training volume by 10%. Day 4: Decrease current training volume by 10%. Day 5: Decrease current training volume by 10%. Day 6: Decrease current training volume by 5%. Day 7: Decrease current training volume by 5%.
  Arms: Taper

SUMMARY:
Purpose: Investigating the effects of stressors and recovery regulation on the super-compensation effect of high-intensity intensive training (IT) in endurance athletes. Methods: This study will recruit 176 competitively trained endurance adult athletes. Participants will conduct a 7-week 3-stage experiment, including 3 weeks of regular training, 3 weeks of 130% progressive IT, and 1 week of 55% taper. Measurement will include training responses (performance and fatigue symptoms), stressors, recovery regulation, and mood state at baseline, during and after regular training, IT, and taper separately. According to the performance after taper, all participants will category into either the responder or non-responder of well-response to supercompensation effect. Statistic analysis: Independent t-test, Chi-squared test, and binary logistic regression will be used to compare the difference in training responses, stressors, recovery regulation, and mood state characteristics between responder and non-responder groups. P value sets at 0.15 for identifying the potential predictors. Logistic stepwise multiple regression will be used further to determine the significant predictors for the responders of well-response to the super-compensation among endurance athletes. P value sets at 0.05.

DETAILED DESCRIPTION:
* Research problems and motivation:

  (1) Research problems: Currently, the primary challenge in sports training monitoring resides in the disparity of responses among athletes to identical high-intensity, high-volume training stimuli (e.g., total distance, frequency, intensity, workload) (Aubry et al., 2015; Aubry et al., 2014; Bellinger, 2020; Le Meur et al., 2014; Le Meur et al., 2013). Despite the widespread dissemination of preventative strategies for overtraining syndrome among coaches and athletes in current sports science research, non-functional overreaching and overtraining syndrome continue to exhibit a prevalence of approximately 19% to 30% in recent years.

  (2) Research motivation: Recent studies have found that following high-intensity, high-volume training, approximately 45.5% to 100% of individuals are categorized as athletes who fail to recover and show poor responses adequately (Aubry et al., 2015; Aubry et al., 2014; Bellenger, Karavirta, et al., 2016; Bellenger et al., 2017; Bellinger, 2020; Fuller et al., 2017; Le Meur et al., 2013; Woods et al., 2018). This phenomenon may be influenced by factors such as inadequate individual recovery capacity or excessive external stressors. Hence, there is an increased emphasis on understanding individual differences, including stressors and recovery regulatory characteristics. By observing the differences between athletes who successfully improve their performance (responders) and those who do not (non-responders) following high-intensity, high-volume training, it may be possible to enhance the precision of future applications of high-intensity, high-volume training in terms of effectiveness and safety.
* Study purpose and hypotheses:

  1. The purpose of this study are two:

     1. To investigate the training responses (sports performance and fatigue symptoms) post-intervention among endurance athletes who exhibit either compensatory training effects (responders) or fail to show such effects (non-responders) following high-intensity, high-volume training. Additionally, it will examine the differences in stressors, recovery regulatory, and emotional state characteristics between these two groups during the intervention period.
     2. To explore the impact of stressors and recovery regulatory characteristics on the presence or absence of compensatory effects following high-intensity, high-volume training among endurance athletes who either respond well or poorly to the intervention. The aim is to understand, through a simple yet comprehensive sideline measurement approach, the characteristics of athletes regarding their ability to adequately recover from fatigue states induced by high-intensity, high-volume training.
  2. The hypotheses of this study:

     1. Endurance athletes who exhibit either compensatory training effects (responders) or fail to show such effects (non-responders) in sports performance are expected to significantly differ in their training responses (sports performance and fatigue symptoms), stressors, recovery regulatory characteristics, and emotional state characteristics.
     2. Certain stressors and recovery regulatory characteristics are expected to have a significant influence on whether endurance athletes exhibit favorable compensatory training effects following high-intensity, high-volume training.
* Study procedure:

  1. Study procedures:

     The study will involve a 7-week experimental protocol divided into 3 phases: 3 weeks of regular training, 3 weeks of gradually increasing high-intensity training at 130%, and 1 week of reduced training at 55% (Bellinger, 2020). Athletes will undergo assessments before, during, and after each phase, including regular training, high-intensity training, and reduced training, to evaluate training responses (sports performance and fatigue symptoms), stressors, recovery regulatory characteristics, and emotional state. Based on athletes' sports performance after the reduced training phase, they will be categorized into two groups: those with favorable compensatory training effects (response group) and those without (non-response group). The detailed weekly training volume design is as follows:

     Stage One: 3 weeks of maintaining participants' regular training habits.

     Stage Two: 3 weeks of high-intensity training (increasing by 10% each week):

     Stage Three: 1 week of reduced training (gradually reduced to 55% of participants' regular training volume): Decrease current training volume followed by 20%, 15%, 10%, 10%, 10%, 5%, and 5% each day.

  (4) Measurement instruments: This study will utilize questionnaires and maximal exercise testing for measurement.
  1. Questionnaire Survey: Participants will be asked to complete the Chinese versions of the Profile of Mood States (POMS) (Hsu, Chang, & Lu, 2003) and the Recovery-Stress Questionnaire for Athletes (RESTQ-Sport) (Chen & Ji, 2002) after each week of training (e.g., every Saturday or Sunday). These questionnaires represent the participants' emotional states and stress-recovery regulatory characteristics. The total questionnaire will be administered 7 times, each session taking approximately 20 minutes.
  2. Maximal exercise testing: Maximal exercise testing will be conducted before and after each stage of the study, including at the beginning of the experiment, after the third week, after the fourth week, after the sixth week, and after the seventh week, totaling 5 maximal exercise tests. Each testing session will take approximately 30 minutes.
* Data collection:

  1. Measurement of Personal Data and Other Relevant Factors:

     1. Personal Data: Before the commencement of the experiment, participants will be asked to complete a personal information form in paper format. This form will record all participants' basic information, including age, height, weight, gender, education level, exercise level, sports specialization, sports performance, medical history, dietary habits, and sleep habits. Additionally, information on risk factors for overtraining syndrome (including exercise performance and fatigue symptoms) and other similar symptomatic diseases (including primary viral diseases, bacterial infections, related inflammatory diseases, diabetes, and hyperthyroidism) will be collected to gather participants' baseline characteristics and exclude overtraining syndrome and other similar symptomatic diseases.
     2. Training Records: During the experiment, all participants' daily training records (including training activities, intensity, and volume) will be electronically recorded to ensure that the expected training intensity is achieved during high-intensity training sessions.
  2. Primary Outcome Measures:

     1. Training response:

        - Performance: This study will conduct progressive maximal exercise tests, including before the experiment starts and after the third, fourth, sixth, and seventh weeks, totaling 5 tests. The results will record participants' resting heart rate, peak power output, maximum heart rate, maximal oxygen uptake, anaerobic threshold, and perceived fatigue index. The tests will be conducted using a progressive resistance cycle ergometer (Corival CPET, LODE, Netherlands). During the test, participants will undergo a 5-minute warm-up at 50 watts with a self-selected pace, followed by a progressive maximal cycle ergometer test. The test will start at 50 watts and increase by 20 watts every minute until the participant cannot maintain a pedaling speed above 10 seconds. After the test, the intensity will be reduced to 50 watts, and participants will pedal at a self-selected pace for 2 minutes, followed by an inquiry about their perceived fatigue index.
     2. Symptom Response:

        * Fatigue Symptoms: Participants will fill out the Chinese version of the Profile of Mood States (POMS) questionnaire after each week's training (e.g., on Sundays), recording their feelings over the past week. The abbreviated Chinese version of the POMS contains 37 mood-related adjectives and takes approximately 3 to 7 minutes to complete. The fatigue subscale score will reflect participants' fatigue symptoms.
        * Emotional State: Participants will complete the Chinese version of the Profile of Mood States (POMS) questionnaire, and the total score for emotional disturbance (= tension + depression + anger + confusion + fatigue - vigor) will be calculated to indicate their overall negative emotional disturbance state.
     3. Stress Recovery Regulation:

        * Stress Sources: Participants will fill out the Chinese version of the Recovery-Stress Questionnaire for Athletes (RESTQ-Sport) after each week's training (e.g., on Sundays), recording their feelings over the past three days. The abbreviated Chinese version of the RESTQ-Sport contains 52 items and takes approximately 15 minutes to complete. General stress and specific sport-related stress scores will reflect participants' stress source characteristics.
        * Recovery Regulation: Participants will complete the Chinese version of the Recovery-Stress Questionnaire for Athletes (RESTQ-Sport), and scores for general recovery and specific sport-related recovery will be calculated to reflect their recovery regulation characteristics.
* Statistical analysis

  1. Firstly, this study will utilize independent t-tests, chi-square tests, and binary logistic regression analyses to compare potential differences between the response (exercise performance and fatigue symptoms), stress sources, recovery regulation, and emotional states of the response and non-response groups. The significance level (P-value) will be set at 0.15.
  2. Secondly, logistic stepwise regression analysis will be employed to identify stress sources and recovery regulation characteristics that significantly influence endurance athletes with or without responses after high-intensity interval training. The significance level (P-value) will be set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Athletes aged 18 or above with endurance-type competitive sports experience. For instance, athletes who have participated in track events of 400 meters or longer, marathons, road cycling, swimming, rowing, race walking, triathlons, orienteering, and similar competitive events.
* A habitual training regimen of at least 6 hours per week. For instance, training three times a week for at least 2 hours each session.
* Minimum of 3 years of training experience, such as being part of a school team or a specialized athlete.
* No severe injuries within the past year. For instance, severe non-regenerative anemia, craniotomy due to cerebral aneurysm, acute myocardial infarction, severe hepatic cirrhosis, severe systemic lupus erythematosus nephritis, severe rheumatoid arthritis, severe head trauma, and similar conditions.
* Not taking substances affecting athletic, physiological, and psychological performance. For instance, unauthorized drugs, prohibited substances, growth hormones like somatotropin and related substances, β2 agonists, hormone and metabolic modulators, diuretics, masking agents, stimulants, anesthetics, cannabis, adrenal corticosteroids, and similar substances.

Exclusion Criteria:

* Presence of an illness resembling symptoms of overtraining syndrome in the week before the start of the experiment. This includes primary viral illnesses, bacterial infections, associated inflammatory diseases, diabetes, or hyperthyroidism.
* Suspected symptoms of high-risk overtraining syndrome in the week preceding the experiment, such as persistent fatigue or exhaustion, unexplained significant decrease in athletic performance exceeding 10%.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 158 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Stressor | Pre-test and the following 7 weeks (follow up once a week)
  The stress score of the recovery-stress questionnaire for athletes (RESTQ-sport) questionnaire.
Recovery regulation | Pre-test and the following 7 weeks (follow up once a week)
  The recovery score of the recovery-stress questionnaire for athletes (RESTQ-sport) questionnaire.
Mood state | Pre-test and the following 7 weeks (follow up once a week)
  The total score of the Profile of Mood State (POMS) questionnaire.
Peak power output | Baseline, the 3rd, 4th, 6th and 7th week
  The peak power output at the end of an incremental exercise test.

SECONDARY OUTCOMES:
Maximal heart rate | Baseline, the 3rd, 4th, 6th and 7th week
  The maximal heart rate at the end of an incremental exercise test.
Fatigue state | Pre-test and the following 7 weeks (follow up once a week)
  The fatigue score of the Profile of Mood State (POMS) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Wun Tsai, Study Chair — Department of Physical Therapy and Assistive Technology, National Yang Ming Chiao Tung University
Locations (1):
- Department of Physical Therapy and Assistive Technology, National Yang Ming Chiao Tung University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steinacker JM, Lormes W, Reissnecker S, Liu Y. New aspects of the hormone and cytokine response to training. Eur J Appl Physiol. 2004 Apr;91(4):382-91. doi: 10.1007/s00421-003-0960-x. Epub 2003 Nov 8. PMID 14608461
- [Background] Meeusen R, Duclos M, Foster C, Fry A, Gleeson M, Nieman D, Raglin J, Rietjens G, Steinacker J, Urhausen A; European College of Sport Science; American College of Sports Medicine. Prevention, diagnosis, and treatment of the overtraining syndrome: joint consensus statement of the European College of Sport Science and the American College of Sports Medicine. Med Sci Sports Exerc. 2013 Jan;45(1):186-205. doi: 10.1249/MSS.0b013e318279a10a. PMID 23247672
- [Background] Matos NF, Winsley RJ, Williams CA. Prevalence of nonfunctional overreaching/overtraining in young English athletes. Med Sci Sports Exerc. 2011 Jul;43(7):1287-94. doi: 10.1249/MSS.0b013e318207f87b. PMID 21131861
- [Background] Cadegiani FA, da Silva PHL, Abrao TCP, Kater CE. Diagnosis of Overtraining Syndrome: Results of the Endocrine and Metabolic Responses on Overtraining Syndrome Study: EROS-DIAGNOSIS. J Sports Med (Hindawi Publ Corp). 2020 Apr 22;2020:3937819. doi: 10.1155/2020/3937819. eCollection 2020. PMID 32373644
- [Background] Halson SL, Jeukendrup AE. Does overtraining exist? An analysis of overreaching and overtraining research. Sports Med. 2004;34(14):967-81. doi: 10.2165/00007256-200434140-00003. PMID 15571428
- [Background] Aubry A, Hausswirth C, Louis J, Coutts AJ, LE Meur Y. Functional overreaching: the key to peak performance during the taper? Med Sci Sports Exerc. 2014 Sep;46(9):1769-77. doi: 10.1249/MSS.0000000000000301. PMID 25134000
- [Background] Aubry A, Hausswirth C, Louis J, Coutts AJ, Buchheit M, Le Meur Y. The Development of Functional Overreaching Is Associated with a Faster Heart Rate Recovery in Endurance Athletes. PLoS One. 2015 Oct 21;10(10):e0139754. doi: 10.1371/journal.pone.0139754. eCollection 2015. PMID 26488766
- [Background] Le Meur Y, Pichon A, Schaal K, Schmitt L, Louis J, Gueneron J, Vidal PP, Hausswirth C. Evidence of parasympathetic hyperactivity in functionally overreached athletes. Med Sci Sports Exerc. 2013 Nov;45(11):2061-71. doi: 10.1249/MSS.0b013e3182980125. PMID 24136138
- [Background] Le Meur Y, Louis J, Aubry A, Gueneron J, Pichon A, Schaal K, Corcuff JB, Hatem SN, Isnard R, Hausswirth C. Maximal exercise limitation in functionally overreached triathletes: role of cardiac adrenergic stimulation. J Appl Physiol (1985). 2014 Aug 1;117(3):214-22. doi: 10.1152/japplphysiol.00191.2014. Epub 2014 Jun 12. PMID 24925979
- [Background] Bellinger P. Functional Overreaching in Endurance Athletes: A Necessity or Cause for Concern? Sports Med. 2020 Jun;50(6):1059-1073. doi: 10.1007/s40279-020-01269-w. PMID 32064575
- [Background] Decroix L, Piacentini MF, Rietjens G, Meeusen R. Monitoring Physical and Cognitive Overload During a Training Camp in Professional Female Cyclists. Int J Sports Physiol Perform. 2016 Oct;11(7):933-939. doi: 10.1123/ijspp.2015-0570. Epub 2016 Aug 24. PMID 26816388
- [Background] Gabbett TJ. The training-injury prevention paradox: should athletes be training smarter and harder? Br J Sports Med. 2016 Mar;50(5):273-80. doi: 10.1136/bjsports-2015-095788. Epub 2016 Jan 12. PMID 26758673
- [Background] Bellenger CR, Karavirta L, Thomson RL, Robertson EY, Davison K, Buckley JD. Contextualizing Parasympathetic Hyperactivity in Functionally Overreached Athletes With Perceptions of Training Tolerance. Int J Sports Physiol Perform. 2016 Jul;11(7):685-92. doi: 10.1123/ijspp.2015-0495. Epub 2015 Dec 1. PMID 26640275
- [Background] Bellenger CR, Thomson RL, Robertson EY, Davison K, Nelson MJ, Karavirta L, Buckley JD. The effect of functional overreaching on parameters of autonomic heart rate regulation. Eur J Appl Physiol. 2017 Mar;117(3):541-550. doi: 10.1007/s00421-017-3549-5. Epub 2017 Feb 11. PMID 28188371
- [Background] Fuller JT, Bellenger CR, Thewlis D, Arnold J, Thomson RL, Tsiros MD, Robertson EY, Buckley JD. Tracking Performance Changes With Running-Stride Variability When Athletes Are Functionally Overreached. Int J Sports Physiol Perform. 2017 Mar;12(3):357-363. doi: 10.1123/ijspp.2015-0618. Epub 2016 Aug 24. PMID 27295717
- [Background] Woods AL, Rice AJ, Garvican-Lewis LA, Wallett AM, Lundy B, Rogers MA, Welvaert M, Halson S, McKune A, Thompson KG. The effects of intensified training on resting metabolic rate (RMR), body composition and performance in trained cyclists. PLoS One. 2018 Feb 14;13(2):e0191644. doi: 10.1371/journal.pone.0191644. eCollection 2018. PMID 29444097
- [Background] Lehmann M, Knizia K, Gastmann U, Petersen KG, Khalaf AN, Bauer S, Kerp L, Keul J. Influence of 6-week, 6 days per week, training on pituitary function in recreational athletes. Br J Sports Med. 1993 Sep;27(3):186-92. doi: 10.1136/bjsm.27.3.186. PMID 8242277
- [Background] Tsigos C, Chrousos GP. Hypothalamic-pituitary-adrenal axis, neuroendocrine factors and stress. J Psychosom Res. 2002 Oct;53(4):865-71. doi: 10.1016/s0022-3999(02)00429-4. PMID 12377295
- [Background] Glass JM, Lyden AK, Petzke F, Stein P, Whalen G, Ambrose K, Chrousos G, Clauw DJ. The effect of brief exercise cessation on pain, fatigue, and mood symptom development in healthy, fit individuals. J Psychosom Res. 2004 Oct;57(4):391-8. doi: 10.1016/j.jpsychores.2004.04.002. PMID 15518675
- [Background] Lakier Smith L. Overtraining, excessive exercise, and altered immunity: is this a T helper-1 versus T helper-2 lymphocyte response? Sports Med. 2003;33(5):347-64. doi: 10.2165/00007256-200333050-00002. PMID 12696983
- [Background] Brooks K, Carter J. Overtraining, Exercise, and Adrenal Insufficiency. J Nov Physiother. 2013 Feb 16;3(125):11717. doi: 10.4172/2165-7025.1000125. PMID 23667795
- [Background] Kreher JB. Diagnosis and prevention of overtraining syndrome: an opinion on education strategies. Open Access J Sports Med. 2016 Sep 8;7:115-22. doi: 10.2147/OAJSM.S91657. eCollection 2016. PMID 27660501
- [Background] Issurin VB. New horizons for the methodology and physiology of training periodization. Sports Med. 2010 Mar 1;40(3):189-206. doi: 10.2165/11319770-000000000-00000. PMID 20199119
- [Background] Costello SE, Rossiter JRW, Howatson G, Bell PG, O'Neill BV, van Someren K, Haskell-Ramsay CF. Effect of intensified training on cognitive function, psychological state & performance in trained cyclists. Eur J Sport Sci. 2023 Jul;23(7):1334-1344. doi: 10.1080/17461391.2022.2097130. Epub 2022 Jul 20. PMID 35771645
- [Background] Dupuy O, Lussier M, Fraser S, Bherer L, Audiffren M, Bosquet L. Effect of overreaching on cognitive performance and related cardiac autonomic control. Scand J Med Sci Sports. 2014 Feb;24(1):234-42. doi: 10.1111/j.1600-0838.2012.01465.x. Epub 2012 Apr 27. PMID 22537000
- [Background] Decroix L, Lamberts RP, Meeusen R. Can the Lamberts and Lambert Submaximal Cycle Test Reflect Overreaching in Professional Cyclists? Int J Sports Physiol Perform. 2018 Jan 1;13(1):23-28. doi: 10.1123/ijspp.2016-0685. Epub 2018 Jan 11. PMID 28422523
- [Background] Hausswirth C, Louis J, Aubry A, Bonnet G, Duffield R, LE Meur Y. Evidence of disturbed sleep and increased illness in overreached endurance athletes. Med Sci Sports Exerc. 2014;46(5):1036-45. doi: 10.1249/MSS.0000000000000177. PMID 24091995
- [Background] Karvonen J, Vuorimaa T. Heart rate and exercise intensity during sports activities. Practical application. Sports Med. 1988 May;5(5):303-11. doi: 10.2165/00007256-198805050-00002. PMID 3387734
- [Background] Hostrup M, Bangsbo J. Limitations in intense exercise performance of athletes - effect of speed endurance training on ion handling and fatigue development. J Physiol. 2017 May 1;595(9):2897-2913. doi: 10.1113/JP273218. Epub 2016 Nov 16. PMID 27673449
- [Background] Manresa-Rocamora A, Flatt AA, Casanova-Lizon A, Ballester-Ferrer JA, Sarabia JM, Vera-Garcia FJ, Moya-Ramon M. Heart rate-based indices to detect parasympathetic hyperactivity in functionally overreached athletes. A meta-analysis. Scand J Med Sci Sports. 2021 Jun;31(6):1164-1182. doi: 10.1111/sms.13932. Epub 2021 Mar 4. PMID 33533045
- [Background] Seggar JF, Pedersen DM, Hawkes NR, McGown C. A measure of stress for athletic performance. Percept Mot Skills. 1997 Feb;84(1):227-36. doi: 10.2466/pms.1997.84.1.227. PMID 9132713
- [Background] Nicholls AR, Backhouse SH, Polman RC, McKenna J. Stressors and affective states among professional rugby union players. Scand J Med Sci Sports. 2009 Feb;19(1):121-8. doi: 10.1111/j.1600-0838.2007.00757.x. Epub 2008 Feb 1. PMID 18248539
- [Background] Roete AJ, Elferink-Gemser MT, Otter RTA, Stoter IK, Lamberts RP. A Systematic Review on Markers of Functional Overreaching in Endurance Athletes. Int J Sports Physiol Perform. 2021 Aug 1;16(8):1065-1073. doi: 10.1123/ijspp.2021-0024. Epub 2021 Jun 8. PMID 34108275
- [Background] Morgan WP, Brown DR, Raglin JS, O'Connor PJ, Ellickson KA. Psychological monitoring of overtraining and staleness. Br J Sports Med. 1987 Sep;21(3):107-14. doi: 10.1136/bjsm.21.3.107. PMID 3676635
- [Background] Raglin JS, Morgan WP, O'Connor PJ. Changes in mood states during training in female and male college swimmers. Int J Sports Med. 1991 Dec;12(6):585-9. doi: 10.1055/s-2007-1024739. PMID 1797703
- [Background] Kellmann M. Preventing overtraining in athletes in high-intensity sports and stress/recovery monitoring. Scand J Med Sci Sports. 2010 Oct;20 Suppl 2:95-102. doi: 10.1111/j.1600-0838.2010.01192.x. PMID 20840567
- [Background] Lastella M, Vincent GE, Duffield R, Roach GD, Halson SL, Heales LJ, Sargent C. Can Sleep Be Used as an Indicator of Overreaching and Overtraining in Athletes? Front Physiol. 2018 Apr 24;9:436. doi: 10.3389/fphys.2018.00436. eCollection 2018. No abstract available. PMID 29740346
- [Background] De Pauw K, Roelands B, Cheung SS, de Geus B, Rietjens G, Meeusen R. Guidelines to classify subject groups in sport-science research. Int J Sports Physiol Perform. 2013 Mar;8(2):111-22. doi: 10.1123/ijspp.8.2.111. PMID 23428482
- [Background] Lochbaum M, Zanatta T, Kirschling D, May E. The Profile of Moods States and Athletic Performance: A Meta-Analysis of Published Studies. Eur J Investig Health Psychol Educ. 2021 Jan 13;11(1):50-70. doi: 10.3390/ejihpe11010005. PMID 34542449
- [Background] Shacham S. A shortened version of the Profile of Mood States. J Pers Assess. 1983 Jun;47(3):305-6. doi: 10.1207/s15327752jpa4703_14. PMID 6886962
- [Background] Morgan WP, Costill DL, Flynn MG, Raglin JS, O'Connor PJ. Mood disturbance following increased training in swimmers. Med Sci Sports Exerc. 1988 Aug;20(4):408-14. doi: 10.1249/00005768-198808000-00014. PMID 3173050
- [Background] O'Connor PJ, Morgan WP, Raglin JS. Psychobiologic effects of 3 d of increased training in female and male swimmers. Med Sci Sports Exerc. 1991 Sep;23(9):1055-61. PMID 1943626
- [Background] Kellmann M, Gunther KD. Changes in stress and recovery in elite rowers during preparation for the Olympic Games. Med Sci Sports Exerc. 2000 Mar;32(3):676-83. doi: 10.1097/00005768-200003000-00019. PMID 10731012
- [Background] Howley ET, Bassett DR Jr, Welch HG. Criteria for maximal oxygen uptake: review and commentary. Med Sci Sports Exerc. 1995 Sep;27(9):1292-301. PMID 8531628